CLINICAL TRIAL: NCT01474044
Title: A Phase IV Study to Evaluate the Efficacy and Safety of Vitamin B12 Contains Extract of Lamb's Stomach in Treatment of Chronic Atrophic Gastritis
Brief Title: To Evaluate the Efficacy and Safety of Vitamin B12 Contains Extract of Lamb's Stomach in Treatment of Chronic Atrophic Gastritis (CAG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinjiang Biochemical Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CATS-CO-002
Record Dates: First submitted 2011-10-27; First posted 2011-11-17 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Atrophic Gastritis (CAG)
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator
- Gastropyloric Complex Capsules (Active Comparator)
  Interventions: Drug: Gastropylor Complex Capsules

INTERVENTIONS:
Drug: Gastropylor Complex Capsules — 3 pills, three times a day, after meal
  Other Names: Gastropyloric Extracts and Vit B12 Complex Capsules
  Arms: Gastropyloric Complex Capsules
Other: Placebo Comparator — Placebo that is same as gastropyloric complex capsules
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Gastropyloric Complex Capsules are safe and effective in the treatment of chronic atrophic gastritis (CAG).

DETAILED DESCRIPTION:
Till now, there is no ideal treatment to chronic atrophic gastritis(CAG). This study is try to find a possible treatment to CAG with Gastropyloric Complex Capsules.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years, male or female
* Histologically diagnosed CAG
* HP negative confirmed by gastric mucosal staining
* Signed an written informed consent

Exclusion Criteria:

* CAG with high-grade intraepithelial neoplasia
* Severe gastric mucosal erosion or bleeding needing treatment
* Active peptic ulcer, GERD, or esophageal stricture
* History of upper GI tract surgery
* History of malignant diseases
* With depression, anxiety neuroses, or hysteria
* Heart failure (NYHA class lll or lV), liver disease (ALT ≥ 80 IU/L, AST ≥ 80 IU/L) or renal disease(Cr ≥ 150 ummol/L)
* Uncontrolled hypertension
* Uncontrolled diabetes
* Alcohol abuse
* Drug allergy
* Participated in another investigational study within 4 weeks prior to Visit 0
* Pregnancy, be a nursing mother or without conception control
* There is any concern by the investigator regarding the safe participation of the participant in the study or for any other reason; the investigator considers the participant inappropriate for participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Effective rate confirmed by histology | within 180 days after treatment
  All patients are required to repeat the histology examination after 180 days follow-up is completed.

SECONDARY OUTCOMES:
clinical manifestations including abdominal pain, anorexia, nausea, vomiting, and belching | within 180 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun WU, Professor, Principal Investigator — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China